CLINICAL TRIAL: NCT03829644
Title: Evaluating the Effects of Six-Week of Lumbar Bracing on Type I Modic Changes: A Pilot Randomised Controlled Trial
Brief Title: Lumbar Bracing for People With Type I Modic Changes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Logistics and Resources
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00086518
Record Dates: First submitted 2019-01-23; First posted 2019-02-04 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain; Bone Marrow Edema; Brace; Modic Changes; Magnetic Resonance Imaging
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, superiority, 1:1 parallel randomised control trial with concealed allocation. Superiority will be based on a minimally clinically significant difference of the Modic changes (our primary outcome measure).
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of each intervention, blinding will not be feasible for participants. However, the MR technician, outcomes assessor, outcome adjudicators, and the statistician will be blinded to the actual allocation. The actual allocation will not be disclosed to the research assistant responsible for image processing, data entry, and the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will be fitted with a semi-rigid prefabricated lumbar brace (Horizon 627 Lumbar Brace, Aspen Medical Company, Oak Canyon, Irvine, CA 92618) in addition to their current back pain management program.
  Interventions: Device: Horizon 627 Lumbar Brace, Aspen Medical Company, Oak Canyon, Irvine, CA 92618
- Control (No Intervention): Participants in this arm will be instructed to follow their current back pain management program.

INTERVENTIONS:
Device: Horizon 627 Lumbar Brace, Aspen Medical Company, Oak Canyon, Irvine, CA 92618 — The brace is an FDA Class I device, one-size adjustable design to fit waists ranging from 24-70 inches. Participants will be instructed to wear the brace for six weeks. As this brace is semi-rigid, it does not prevent motion - only reduces motion in the lumbar areas. Our prior work and that of others have shown that this type of bracing does not reduce spinal function and is not associated with atrophy.
  Arms: Intervention

SUMMARY:
Despite the high prevalence of low back pain, little is still known about its underlying pathology. Only a small proportion of people (~1%) have a diagnosable pathoanatomical entity causing low back pain. The other types of back pain are classified as non-specific low back pain. Thus, current back pain management typically focuses on relieving symptoms. This is largely ineffective without understanding the cause. Yet, there are some pathologies which are thought to be associated with low back pain.

Vertebral bone marrow oedemas are now known to be a hallmark feature for low back pain. There are three types of vertebral bone marrow oedemas. Type I oedemas are dynamic lesions that may progress to a higher grade, stop, or even return to normal. Although the precise cause of type I oedemas is not well understood, loading on the spine plays a key role in its development. Lumbar braces are known to reduce loads on the spine. Thus, they may reduce the size of oedema by modifying loads on the spine. The investigators already know that wearing a lumbar brace reduces pain in people with back pain and type I vertebral bone marrow oedemas. Unfortunately, there is no study showing that pain reduction with bracing is associated with a reduction of oedema. The goal of this study is to determine if wearing a lumbar brace for six weeks will reduce the dimensions of type I vertebral bone marrow oedema.

DETAILED DESCRIPTION:
Purpose

Modic changes are now known to have a high specificity for low back pain. Modic changes represent bone oedema and are dynamic lesions that may progress to a higher grade, stop, or even reverse to a lower grade. Although the precise aetiology of Modic changes is not well understood currently, abnormal mechanical loading plays a key role in their development and progression. Biomechanical studies have demonstrated that abnormal shear forces acting on the vertebral endplate could lead to endplate microtrauma and marrow oedema correlating with type I Modic changes. This suggests that Modic changes may be ideal structural targets for treatment designed to alter vertebral loading. The main goal of this project is, therefore, to mitigate, stop, or reverse Modic lesion progression and their associated pain through the use of lumbar orthoses that can modify loads acting on the lumbar spine by limiting both fine and gross trunk movements, and thus decreasing demands for muscular activities. As this effect of bracing likely reduces biomechanical stress on the vertebral endplate as well, lumbar orthoses should, in theory, be able to impact bone marrow lesions by normalizing lumbar loading.

Hypothesis

I) Modification of the mechanical load in the lumbar spine using a semi-rigid lumbosacral orthosis for six weeks will reduce the dimensions of Modic changes

II) The same bracing protocol will help mitigate, stop, or reverse the progression of Modic changes;

III) These morphologic changes will be associated secondarily with a reduction in pain and discomfort and an increase in spinal function.

Although the precise aetiology of Modic changes is not well understood, abnormal mechanical loading likely plays an important role in their development and progression. Biomechanical studies have demonstrated that abnormal shear forces acting on the vertebral endplate could lead to endplate microtrauma and marrow oedema correlating with type I Modic changes. Modic changes are dynamic lesions that may progress to a higher grade, stop, or even reverse to a lower grade. All of this suggests that Modic changes may be ideal structural targets for treatment that can alter vertebral loading.

Objectives

I) PRIMARY: To determine if wearing a semi-rigid lumbosacral orthosis for six weeks will significantly reduce the dimensions of Modic changes;

II) SECONDARY: To determine if this same bracing protocol will induce morphological and textural changes in the vertebra;

III) SECONDARY: To determine if these changes are associated with improvements in pain and function;

IV) EXPLORATORY: To determine if this same bracing protocol will reduce prescription and/or consumption of analgesics;

V) EXPLORATORY: To determine if this same bracing protocol will reduce the low back pain related use of health resources.

Methods/Procedures

This project is a prospective, superiority, 1:1 parallel randomised control trial with concealed allocation. Randomisation arms include semi-rigid lumbar bracing and no bracing. Superiority will be based on a minimally clinically significant difference of the Modic changes (our primary outcome measure).

After obtaining approval from the University of Alberta's Health Research Ethics Board, the investigators will invite 46 volunteers with benign low back pain and MRI evidence of type I Modic changes to consent and participate in this study. the investigators will recruit volunteers from the University of Alberta Hospital who have obtained clinical MRIs in their regular course of care who have been identified as having a Modic change in their lumbar spine.

A co-investigator will review all routine lumbar spine MR images from the Department of Radiology of the University of Alberta to identify possible participants who have been identified as having a Modic change as part of their usual clinical care (a waiver for consent will be requested in this application). A letter of invitation will then be sent to those persons inviting them to contact us for more information about the study. A research assistant will respond to all inquiries and then administer the Numeric Pain Rating Scale and the Oswestry Disability Index to further screen the participants for minimal score values to prevent floor effects of outcome response. If potential participants meet these inclusion criteria and provide written informed consent, the research coordinator will enrol them in the study.

After enrolment, each participant will be given a study number to maintain and track her/his records. The participant will be then provided with a Research Electronic Data Capture (REDCap) secure web address to complete various data collection surveys (e.g. demographics).

All participants will be instructed that the current study will not substitute their current back pain management program. Participants in the intervention arm will be fitted with a semi-rigid prefabricated lumbar brace (Horizon 627 Lumbar Brace, Aspen Medical Company, Oak Canyon, Irvine, CA 92618). The brace is a one-size adjustable design to fit waists ranging from 24-70 inches. Participants will be instructed to wear the brace for six weeks. As this brace is semi-rigid, it does not prevent motion - only reduces motion in the lumbar areas. Our prior work and that of others have shown that this type of bracing does not reduce spinal function and is not associated with atrophy.

Baseline session

The investigators will collect demographics (e.g., age, sex, family physician contact), previous history/comorbidities, past imaging, and current treatment. As the initial MR images used to identify potential participants may be taken for proposes other than visualizing Modic changes, their quality may not be appropriate for quantitative image processing. Therefore, all participants will undergo baseline MR imaging. Imaging protocols for the sagittal T2-weighted scans will be as follows: position: supine; repetition time: 1960 ms; echo time: 106 ms, slice thickness:4.0 mm; and matrix size:512×512. Likewise, the anticipated MRI parameters for the fast spin-echo sagittal T1-weighted scans will be as follows: position: supine; repetition time: 340 ms; echo time: 12.9 ms; slice thickness: 4.0 mm and matrix:512×512. The sequences and timings will be kept consistent across all participants.

The investigators will randomise participants to one of two arms: semi-rigid lumbosacral orthosis or no brace following imaging to confirm the presence of Modic changes in these new images.

Randomisation

The investigators will deploy the REDCap randomisation tool to assign participants evenly into the intervention and control groups. The tool uses a defined parameter (subject ID in this study) to create a template allocation table. The on-site research assistant will enter each participant's REDCap record and then click the "Randomize" button. This will trigger REDCap to check the allocation table and display the group to which the participant should be assigned. The assignment is permanent and not editable within the participant record and, like all other activity within REDCap, is tracked and not modifiable in the audit log.

MR imaging

After enrollment, all subsequent imaging will be carried out at the MRI Research Center at Edmonton's Cross Cancer Institute using a 3T whole-body Philips MRI scanner (Philips Healthcare Intera). Based on a previous study, the anticipated MRI parameters for the sagittal T2-weighted scans will be as follows: position: supine; repetition time: 1960 ms; echo time: 106 ms, slice thickness:4.0 mm; and matrix size:512×512. Likewise, the anticipated MRI parameters for the fast spin-echo sagittal T1-weighted scans will be as follows: position: supine; repetition time: 340 ms; echo time: 12.9 ms; slice thickness: 4.0 mm and matrix:512×512. The sequences and timings will be kept consistent across all participants.

Self-reported questionnaires

The investigators will measure participants' pain level using the Numeric Pain Rating Scale. The investigators will use the Roland-Morris Disability Questionnaire and the Oswestry Disability Index to measure participant function and disability level.

Immediately after wearing the brace (only the intervention group)

To assess the immediate impact of the brace, participants will use self-reported outcome tools on the REDCap to quantify pain (Numeric Pain Rating Scale) immediately after wearing the brace.

To measure the quality (how tightly the brace has been worn) and quantity (how much time the brace has been worn) of brace usage, a low-powered portable heat and load monitoring system will be embedded within the pressure pad of the brace. The force measurement part of the monitoring system is sensitive to the forces normal to the brace surface, but not to shear forces, and can be deployed to monitor the quality of the brace wear by participants.28 The temperature part of the monitoring system gives an accurate and stable output over the temperature range from 5 °C to 50 °C,29 and can be deployed to monitor how long the brace has been worn during the brace treatment.

Weeks 1 to 6 follow-ups

All participants will receive a series of text questions by mobile phone 3 times a week for 6 weeks. The questions will collect data related to the pain (Numeric Pain Rating Scale), spinal function (Roland-Morris Disability Questionnaire and Oswestry Disability Index), brace usage, and analgesic consumption.

Week 6 MRI scanning

At this visit, the investigators will administer the Numeric Pain Rating Scale, Oswestry Disability Index, and self-reported Roland-Morris Disability Questionnaire. All participants will then undergo a follow-up MRI scan using the very MR imaging protocol.

The costs of the first and second MRI will be paid by a grant from the Alberta Spine Foundation. The investigators will not use the clinical images taken at the designated centres in this study. These initial clinical images are only used for Dr. Dhillon to identify potential participants. The investigators will not use them further in our study as their specific parameters vary too much to be used in our study.

Week 7 to 52 follow-ups

The investigators will continue to collect a series of outcomes and interview questions (Numeric Pain Rating Scale, Roland-Morris Disability Questionnaire, Oswestry Disability Index, brace usage, and analgesic consumption), by short message service at 4, 8 and 12 months.

End of the enrollment

The investigators will use participant personal health numbers (obtained at baseline with consent) to perform an exploratory analysis through the Alberta Bone and Joint Health Network of health care resource utilization in the year before and during the trial (e.g. prescriptions filled, primary care and emergency department visits, imaging usage, etc.).

Image and Data Analysis

Blinding

Due to the nature of each intervention, blinding will not be feasible for participants. However, the MR technician, outcomes assessor, outcome adjudicators, and the statistician will be blinded to the actual allocation. The actual allocation will not be disclosed to the research assistant responsible for image processing, data entry, and the statistician. The investigators will develop two interpretations of our results based on a blinded review of the primary outcome data (intervention A vs. intervention B). One scenario will assume intervention A was brace and the other will assume intervention A was routine recommendations. Only after our team has agreed that there will be no further changes in the interpretation of the scenarios will the randomisation code be broken, and the correct interpretation used in manuscript preparation.

Image analysis and processing

Image processing will be carried out offline using highly reliable Matlab®-based (MathWorks, Natick, MA) lumbar spine analysis software for MRI images developed by our team. The software uses signal and textural variations in the neighbouring structures to semi-automatically segment vertebrae and intervertebral discs from adjacent tissues. It then calculates traditional measures such as mean signal intensity, area, disc height, width, the range of signal intensity as well as more than two hundred textural features, including kurtosis, skewness, contrast, homogeneity, energy, and correlation for each region of interest.

Statistical Analysis

The investigators will employ a repeated measure ANOVA to compare pain level between groups. The investigators will use age, gender, brace type, and pain severity as potential covariates if randomisation does not result in group equivalence. The investigators will also estimate the effect size of differences between and within the groups for pain using Cohen's d.

ELIGIBILITY:
Inclusion Criteria:

* Pain between the 12th rib and buttocks with or without symptoms into one or both legs, which, in the opinion of the examiner, originate from the lumbar region
* Have MRI evidence of type I Modic changes
* Have a baseline Oswestry Disability Index >25%
* Aged between 18 and 65 years
* Are ambulatory
* Can read and understand English
* Living in Edmonton, Alberta, Canada

Exclusion Criteria:

* Back pain due to a systemic or specific disease such as known cancer, spinal infection, fracture, or ankylosing spondylitis
* Severe pain in the hip and knee joints
* Claustrophobia
* Any contraindications for MRI, such as pacemakers, orthopaedic prosthesis, device or implants at the spine or pelvic girdle
* Pregnancy
* Implanted with an intrauterine contraceptive device
* Significant compression of the spinal cord/nerves
* Previous back surgery
* Waist circumference greater than 70 inches
* Have received back injections within the last 4 weeks
* On-going workers' compensation or litigation cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change in the pain level | Week 6
  Change in the pain level between the baseline and 6-week follow-up will be evaluated using the Numeric Pain Rating Scale [0-10].
Change in the pain level | Month 4
  Change in the pain level between the baseline and 4-month follow-up will be evaluated using the Numeric Pain Rating Scale [0-10].
Change in the pain level | Month 8
  Change in the pain level between the baseline and 8-month follow-up will be evaluated using the Numeric Pain Rating Scale [0-10].
Change in the pain level | Month 12
  Change in the pain level between the baseline and 12-month follow-up will be evaluated using the Numeric Pain Rating Scale [0-10].
Change in the size of the bone marrow lesions | Week 6
  Change in the size of the bone marrow lesion (Modic Changes) between the baseline and six-week follow-up will be evaluated by measuring the area of the lesion.
Change in the size of the texture of marrow lesions | Weeks 0 and 6
  Change in the texture of the bone marrow lesion (Modic Changes) between the baseline and six weeks will be evaluated using grey level co-occurrence matrix (Contrast, correlation, homogeneity, and the entropy).

SECONDARY OUTCOMES:
Change in the self-reported Disability Level - Questionnaire A | 6 Weeks
  Change in the self-reported disability between the baseline and 6-week follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported Disability Level - Questionnaire A | 4 Months
  Change in the self-reported disability between the baseline and 4-month follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported Disability Level - Questionnaire A | 8 Months
  Change in the self-reported disability between the baseline and 8-month follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported Disability Level - Questionnaire A | 12 Months
  Change in the self-reported disability between the baseline and 12-month follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported Disability Level - Questionnaire B | 6 weeks
  Change in the self-reported disability between the baseline and 6-week follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale].
Change in the self-reported Disability Level - Questionnaire B | 4 months
  Change in the self-reported disability between the baseline and 4-month follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale].
Change in the self-reported Disability Level - Questionnaire B | 8 months
  Change in the self-reported disability between the baseline and 8-month follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale].
Change in the self-reported Disability Level - Questionnaire B | 12 months
  Change in the self-reported disability between the baseline and 12-month follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale] between.

OTHER OUTCOMES:
Change in healthcare resource utilization- regulated prescriptions filled (after enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related regulated prescriptions filled from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- primary care visits (after enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related primary care visits from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- specialist visits (after enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related specialist visits from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- imaging (after enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related imaging from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- allied health visits (after enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related allied health visits from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- regulated prescriptions filled (before enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related regulated prescriptions filled from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- primary care visits (before enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related primary care visits from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- specialist visits (before enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related specialist visits from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- imaging (before enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related imaging from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- allied health visits (before enrollment) | 12 months
  The change in healthcare resource utilization, measured by counting the number of back-pain related allied health visits from the past 12 months before enrollment and baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Kawchuk, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No